CLINICAL TRIAL: NCT06066749
Title: Efficacy of Respiratory Protection Against the Effects of Wood Smoke Exposure in Young Healthy Adults
Acronym: MASKON
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: MASKON has been suspended while the study activities are transferred from the EPA Human Studies Facility in Chapel Hill to the EPA Office of Research and Development headquarters at Research Triangle Park.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-1135
Record Dates: First submitted 2023-09-18; First posted 2023-10-04 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Wood Smoke; Respirators; Masking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wood Smoke 1 (Experimental): Volunteers will be be exposed to woodsmoke for 2 hours while exercising in specialized exposure chamber. Woodsmoke (WS) will be generated by smoldering untreated oak and diluting the resulting WS emissions with clean air to achieve a target concentration of WS in the exposure chamber at an average of approximately 500 μg/m3 for the 2-hour exposure period. During the exposure, participants will exercise intermittently using a stationary bicycle with rest periods (i.e., 4 x 15 minutes on, 4 x 15 minutes off). The workload on the bicycle will be pre-determined on the training day to produce a minute ventilation rate of approximately 25 L/min/m2, which is considered a moderate level of exercise.
  Interventions: Other: Filtration of all PM and VOC's; Other: Filtration of VOC's

INTERVENTIONS:
Other: Filtration of all PM and VOC's — During each exposure session, participants will wear a modified MaxAIR controlled air pressure respirator (CAPR) manufactured by Syntech International (BMD), Irvine, CA, USA, that will deliver filtered woodsmoke directly to the participant. The MaxAIR CAPR is a NIOSH approved (TC 21C-1050) powered air purifying respirator used for infectious disease control in laboratory and medical settings.
  In the modified MAXAIR CAPR used during this study's exposure sessions, an external pump and different filtering media. For this intervention, virtually all particulate matter (PM) and volatile organic compounds (VOC's) will be removed using commercially available P100/VOC respirator filters (3M cartridge; 60925 or equivalent).
Other: Filtration of VOC's — During each exposure session, participants will wear a modified MaxAIR controlled air pressure respirator (CAPR) manufactured by Syntech International (BMD), Irvine, CA, USA, that will deliver filtered woodsmoke directly to the participant. The MaxAIR CAPR is a NIOSH approved (TC 21C-1050) powered air purifying respirator used for infectious disease control in laboratory and medical settings.
  In the modified MAXAIR CAPR used during this study's exposure sessions, an external pump and different filtering media. For this intervention, virtually all particulate matter (PM)will be removed using commercially available P100 respirator filters (DM; cat. # 2097).

SUMMARY:
Purpose: This study is designed to test whether the gaseous fraction of woodsmoke, volatile organic compounds, produce acute cardiac, respiratory, and systemic inflammatory health effects after controlled exposure to woodsmoke in health, young volunteers.

Participants: Approximately fifty, 18-35 year-old healthy volunteers to complete the study.

Procedure: After consenting to participate in the study, participants will undergo two exposures to approximately 500 μg/m3 woodsmoke. The two exposures will be held at least 3 weeks apart. Each exposure session will have a follow-up session approximately 24 hr later. During each exposure session, participants will wear a modified MAXAir Systems (Irvine, CA, USA) (TC 21C-1050) controlled air pressure respirator (CAPR) that will deliver filtered woodsmoke directly to the participant's breathing zone. During the first exposure, the CAPR will deliver woodsmoke from which virtually all particulate matter (PM) and volatile organic compounds (VOC's) will be removed. During the second exposure, only the PM will be removed from the woodsmoke, allowing the VOC to pass into the subject's breathing zone. During each session, participants will be exposed for 2 hours while exercising intermittently (15 min exercise followed by 15 min rest) on a stationary bike at a workload sufficient to maintain a minute ventilation of approximately 25 L/min/m2. Venous blood samples and measurements of respiratory, cardiac, and vascular function will be performed prior, immediately following and approximately 18 hrs post each exposure. Approximately 24 hours post-exposure, participants will undergo a bronchoscopy procedure to sample bronchoalveolar fluid and cells for evidence of an inflammatory response to the exposures. Nasal epithelial lining fluid will be also collected approximately 24 hours post each exposure.

DETAILED DESCRIPTION:
Wood smoke pollution is a common problem across the world, including in the US. This wood smoke comes from people using wood to heat and cook, as well as from wildfires. Woodsmoke (WS) derived from wildland fires account for a significant fraction of ambient air pollution, including particulate matter (PM) and volatile organic compounds (VOCs) in the gaseous phase. It remains unclear whether the gaseous fraction of woodsmoke contributes to acute or chronic health effects. The present study is designed to test whether the gaseous fraction of woodsmoke, volatile organic compounds, produce acute cardiac, respiratory, and systemic inflammatory health effects after controlled exposure to woodsmoke in health, young volunteers. Results from this study will also increase understanding of how wood smoke exposure adversely affects the functioning of the human cardiovascular and respiratory systems. This understanding may be especially important for patients with cardiopulmonary diseases.

Study design Volunteers will participate in two exposure sessions. Each exposure session will be 2 hours in duration and will take place in a specialized exposure chamber. Woodsmoke (WS) will be generated by smoldering untreated oak and diluting the resulting WS emissions with clean air to achieve a target concentration of WS in the exposure chamber at an average of approximately 500 μg/m3 for the 2-hour exposure period. During the exposure, participants will exercise intermittently using a stationary bicycle with rest periods (i.e., 4 x 15 minutes on, 4 x 15 minutes off). The workload on the bicycle will be pre-determined on the training day to produce a minute ventilation rate of approximately 25 L/min/m2, which is considered a moderate level of exercise. During the exposure, fluctuations in the WS concentration will be corrected by controlling the flow of dilution air. The concentrations of carbon monoxide and nitrogen oxides will be monitored continuously to maintain the safety of the atmosphere.

During each exposure session, participants will wear a modified MaxAIR controlled air pressure respirator (CAPR) manufactured by Syntech International (BMD), Irvine, CA, USA, that will deliver filtered woodsmoke directly to the participant. The MaxAIR CAPR is a NIOSH approved (TC 21C-1050) powered air purifying respirator used for infectious disease control in laboratory and medical settings. The CAPR is a commercially available, integrated helmet system that delivers filtered air directly to the participant's breathing zone. A flexible lens (shield) with a thin film cuff is attached to the front of the helmet. The thin filament is pulled under the participant's chin to ensure that breathing space is enclosed but not sealed. This allows air to "leak" around the cuffs margin using positive pressure generated by the internal air pump.

In the modified MAXAIR CAPR used during this study's exposure sessions, an external pump and different filtering media will be added to remove volatile organic compounds and/or particulate matter from the woodsmoke being delivered to the breathing space. The flow rate generated will be significantly higher than the participant's maximum peak inspiratory flow to ensure a positive pressure is maintained during the entire two-hour exposure session. Additional safety monitoring enhancements, notably a pressure sensor at the interface of the tubing bundle and pump heads, have been added to ensure that the pump maintains a constant flow and pressure as it delivers filtered woodsmoke to the volunteer's breathing zone.

During one of the exposures, virtually all particulate matter (PM) and volatile organic compounds (VOC's) will be removed using commercially available P100/VOC respirator filters. During the other exposure, only the PM will be removed from the woodsmoke. The participant will be blinded as to what filters are used during each exposure. The flow rate of filtered woodsmoke into the CAPR will be monitored to ensure that it exceeds the respiratory rate and peak inspiration flow of the subject (>180 lpm). The PM filtering medium used with this respirator will be P100 filters (3M, cat. #: 2097) or equivalent. The PM/VOC filter will consist of 3M cartridge (60925 or equivalent). A follow-up visit will be scheduled approximately 24 hr after each exposure during which bronchoalveolar lavage and NELF procedures will be performed (as described below).

ELIGIBILITY:
Inclusion criteria

1. Age 18-35 years old, healthy individuals (Body Mass Index (BMI, kg/m2) values ≥ 19 and ≤ 34, inclusive).
2. Weight equal to or greater than 110 lbs. (Requirement to complete bronchoscopy procedure)
3. Physical conditioning that allows intermittent, moderate exercise for approximately 60 min during a 2-hour exposure session. The volunteer must be able to complete the exposure exercise regimen at a workload sufficient to induce a minute ventilation rate of approximately 25 L/min/m2 for 15 min without exceeding 80% of projected maximal heart rate.
4. Normal ECG.
5. Normal lung function based on NHANES III reference values: Forced vital capacity (FVC) ≥ 80% of that predicted for age, gender, ethnicity, and height; Forced expiratory volume in one second (FEV1) ≥ 80% of that predicted for age, gender, ethnicity, and height; FEV1/FVC ratio ≥ 70% (absolute value).
6. Oxygen saturation greater than 94% at the time of physical exam.

Exclusion criteria

1. Individuals with the following conditions: a) A history of acute or chronic cardiovascular disease, chronic respiratory disease, cancer, rheumatologic disease, neuromuscular disease, or immunodeficiency state, b) Blood pressure readings ≥ 140 systolic and/or ≥ 90 diastolic, c) Diabetes (previously diagnosed or with hemoglobin A1c level equal to or greater than 6.4%) d) Asthma or a history of asthma, e) Bleeding/clotting disorders.
2. Individuals with a cardiovascular disease risk score greater than 10% using the ACC/AHA ASCVD risk calculator. (Based on the 10-year risk of heart disease or stroke using the Atherosclerotic Cardiovascular Disease algorithm published in 2013 American College of Cardiology/American Heart Association Guideline on the Assessment of Cardiovascular risk.)
3. Individuals who have unspecified illnesses, which in the judgment of the medical staff might increase the risk associated with woodsmoke inhalation will be a basis for exclusion.
4. Individuals who have had recent (within 6 month) abdominal and/or eye surgery, or with any types of hernia, as well as any other contraindications for raised intra-abdominal pressure.
5. Individuals who are currently taking systemic steroids or oral anticoagulants long term.
6. Individuals who are taking prescribed medications such as ß-blocker medications, that may impact the results for the duration of the study. Other medications not specifically mentioned here may be reviewed by the medical staff prior to an individual's inclusion in the study. Use of other medications will be evaluated on a case-by-case basis. There is the potential that an individual's current medication use will preclude them from participating in the study at the current time, but they may be reassessed and potentially rescheduled for participation later based on the judgement of the medical staff.
7. Individuals who are allergic to:

   * Chemical vapors or gases.
   * Tape or electrodes on their skin.
   * Or individuals with active allergies or currently experience allergy related symptoms
8. Individuals who are pregnant, attempting to become pregnant or breastfeeding.
9. Individuals who are currently smoking (including vaping, hookah and e-cigarette) or have smoking history within 1 year of study or have an equal to greater than or a 5-pack year smoking history.
10. Individuals living with a smoker who smokes inside the house.
11. Individuals who are regularly exposed to high levels of vapors, dust, gases, or fumes.
12. Individuals who do not read, speak, or understand English well enough to give informed consent.
13. Individuals that are unable to perform the exercise required for the study.
14. Individuals who are unwilling or unable to stop taking any current dietary supplements or vitamins for the duration of the study.
15. Individuals currently taking Omega-3 supplements (i.e. fish oil, krill oil, algae oil).
16. Individuals currently taking prebiotics, probiotics, or antihistamines.
17. Individuals who have experienced an acute respiratory illness within the last 6 weeks.
18. Individuals who have a facial hair or hair style that will interfere with the CAPR seal based on the study team's assessment.
19. Individuals with allergies to the medications used in the bronchoscopy procedure.
20. Individuals with a naris that is too restrictive to permit the fiberoptic bronchoscope to pass comfortably.
21. Regular use of cromolyn (except for prophylaxis of exercise induced bronchospasm) or any use of leukotriene inhibitors (Montelukast or Zafirlukast) within the past month.
22. Night-time symptoms of cough or wheezing greater than 1x/week.
23. Regular use of aspirin or other nonsteroidal anti-inflammatory drug (which inhibit platelet function).
24. Individuals who are not willing to comply with the following requirements: a) Avoid smoke and fumes for 24 hours before all visits, b) Avoid dusty and smoky places for 48 hours prior to follow-up visit, c) Cannot take anything by mouth after midnight the day of the bronchoscopy, d) Cannot travel by bike or motorcycle for any study visit, e) Cannot travel out of town for 24 hours after bronchoscopy, f) Avoid exposure to unvented household combustion sources (gas stoves, lit fireplaces oil/kerosene heaters) for 48 hours before all visit, g) Cannot take any prescription or over-the-counter medications (excluding birth control) for one-week prior to bronchoscopy, h) Avoid drinking alcohol 24 hours before all visits, i) Avoid strenuous exercise for 24 hours prior to and after all visits, j) Eat a light breakfast and low-fat lunch on the exposure day, k) Refrain from eating pan fried and/or grilled foods 12 hours prior to the exposure days, l) Refrain from consuming caffeine for 12 hours prior to all study visits, m) Refrain from consuming food 2 hours prior to the consenting and follow up sessions, as this may interfere with induced sputum collection, n) Wear a N95 mask during all visits to the HSF. A mask will be provided for you upon check-in to the facility, o) Arrive to the medical station within 15 minutes of their scheduled visit time.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in polymorphonuclear neutrophils (PMN%) in the Bronchoalveolar lavage fluid (BAL) | Approximately 24 hours post exposure.
  Airway inflammation will be assessed by the % PMN in the (BAL)

SECONDARY OUTCOMES:
Change in Forced Expired Volume in the First Second (FEV1) (liter) | Immediately after each exposure and approximately 24 hours post exposure.
  FEV1 is determined by spirometry
Change in Forced Vital Capacity (FVC) (liter) | Immediately after each exposure and approximately 24 hours post exposure.
  FVC is determined by spirometry
Change in Diameters (mm) of Retinal Arteries and Veins | Immediately after each exposure and approximately 24 hours post exposure.
  Retinal images will be taken using an FDA-approved, commercially available, non-mydriatic fundus camera. Images will be taken from both eyes.
Percent Change in Heart Rate Variability | Immediately after each exposure and approximately 24 hours post exposure.
  Heart rate variability will be collected by the Holter monitor recording.
Change in concentration of Blood Fatty Acids (ng/mL) | Immediately after each exposure and approximately 24 hours post exposure.
  Blood sample will be collected for fatty acids analysis.
Change in concentration of Blood Cholesterol (ng/mL) | Immediately after each exposure and approximately 24 hours post exposure.
  Blood sample will be collected for blood cholesterol analysis.
Change in concentration of Cytokines in Nasal Epithelial Lining Fluid (NELF) (ng/mL) | Immediately after each exposure and approximately 24 hours post exposure.
  NELF samples will be collected for cytokine measurements.
Change in concentration of interleukin-6, interleukin-8, interleukin-1 beta, and tumor-necrosis factor alpha in blood. (pg/mL) | Immediately after each exposure and approximately 24 hours post exposure.
  Blood will be collected prior to and post exposure to analyze for inflammatory markers.
Change in concentration of C-reactive protein in blood. | Immediately after each exposure and approximately 24 hours post exposure.
  Blood will be collected prior to and post exposure to analyze for inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: James Samet, Principal Investigator — Environmental Protection Agency (EPA)
Locations (1):
- U.S. Environmental Protection Agency Human Studies Facility, Chapel Hill, North Carolina, United States